CLINICAL TRIAL: NCT05758324
Title: Prospective, Randomized, Double-blind, Parallel-group Study Evaluating the Effect of a Specific Trace Metal Complex Versus Placebo on the Severity of Apnea in Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Study Evaluating the Effect of a Specific Trace Metal Complex Versus Placebo on the Severity of Apnea in Patients With Obstructive Sleep Apnea Syndrome
Acronym: OLIGO-SAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratoires Pronutri (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-A01340-43
Record Dates: First submitted 2023-02-19; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Apnea, Obstructive
Keywords: trace elements; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trace elements (Experimental): Nutri PNEA in a single dose (4 sequences of 10 tablets). Nutri PNEA is a complex of trace elements with the status of a food supplement.
  Interventions: Dietary Supplement: Nutri PNEA
- Placebo (Placebo Comparator): 4 sequences of 10 tablets containing only excipients
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutri PNEA — 4 sequences of 10 tablets (one intake)
  Arms: Trace elements
Dietary Supplement: Placebo — 4 sequences of 10 tablets (one intake)
  Arms: Placebo

SUMMARY:
Obstructive sleep apnea syndrome (OSA) is defined by the association of clinical symptoms - drowsiness in particular - and sleep breathing disorders, objectified by measuring the apnea-hypopnea index (AHI). Apneas and hypopneas during sleep are responsible for micro-arousals and hypoxemia.

In the short term, these result in daytime sleepiness with reduced alertness, difficulty driving and carrying out tasks (increased risk of road accidents and accidents at work), memory and concentration problems. , mood disorders. These disturbances lead to an impairment of the quality of life.

In the long term, severe OSA (AHI > 30 events/hour) increases all-cause mortality and cardiovascular morbidity.

The reference treatment is nasal ventilation by Continuous Positive Airway Pressure (CPAP). In practice, the observance and effectiveness of CPAP are limited by the sometimes difficult acceptance of cumbersome equipment, involving noise pollution and requiring the wearing of night-time equipment that some patients find difficult to bear.

The alternative treatment is represented by the mandibular advancement orthosis . Lifestyle and dietary measures are always recommended.

To date, no pharmacological treatment has demonstrated its effectiveness in OSA.

Studies have shown that the antioxidant capacity of the blood is reduced in patients with OSA. It would be secondary to the cycles of hypoxia and reoxygenation which cause a modification of the oxidative balance, leading to an increase in free radicals. It has been observed that the serum levels of trace elements and heavy metals are higher during OSA, by deterioration of the balance of these substances due to oxidative stress and inflammation.

Antioxidant therapies have reduced biomarkers of oxidative stress in apneic patients.

A new path of research is opening up with the use of antioxidants and trace elements in OSA.

To scientifically support the hypothesis of the action of these supplements based on trace metals on OSA, PRONUTRI wish to conduct a comparative, randomized, double-blind study versus placebo evaluating the effect of a specific complex of trace metals in the OSA.

ELIGIBILITY:
Inclusion Criteria:

* adult patient with moderate to severe sleep apnea-hypopnea syndrome confirmed by polysomnography dating less than 3 months with an apneas/hypopneas index ≥ 15 events/h
* stable weight (5% variation of the weight at the time of the polysomnography done within 3 months)

Exclusion Criteria:

* patient previously treated for OSA by continuous positive airway pressure or mandibular orthosis
* obesity (body mass index > 30 kg/m2)
* pregnant or post-pregnancy women less than 6 months old or of childbearing age without an effective method of contraception
* respiratory, cardiac, hepatic or renal failure
* active cancer or history of cancer
* alcohol abuse
* antidepressant intake
* use of compression stockings
* intake of product or supplementation enriched with trace metals and/or trace elements and/or mineral salts and/or vitamins.
* taking any type of psychotropic medication
* previous intake of trace elements to treat OSA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of apneas/hypopneas | 60 days

SECONDARY OUTCOMES:
Change in Ventilatory Response | 60 days
  Change in Ventilatory Response assessed by tests of Ventilatory Response to Carbon Dioxide (CO2)
Proportion of patients with a 50% reduction in the apnea-hypopnea index | 60 days
  AHI is used to diagnose obstructive sleep apnea by counting respiratory events. An index greater than 5 per hour defines a ventilatory disorder.
  AHI defines severity as well, the index is:
  Mild, between 5 and 15 per hour Moderate, between 15 and 30 per hour Severe, over than 30 per hour
Proportion of patients with an apnea-hypopnea index < 30/hour | 60 days
  AHI is used to diagnose obstructive sleep apnea by counting respiratory events. An index greater than 5 per hour defines a ventilatory disorder.
  AHI defines severity as well, the index is:
  Mild, between 5 and 15 per hour Moderate, between 15 and 30 per hour Severe, over than 30 per hour
Proportion of patients with an apnea-hypopnea index < 15/hour | 60 days
  AHI is used to diagnose obstructive sleep apnea by counting respiratory events. An index greater than 5 per hour defines a ventilatory disorder.
  AHI defines severity as well, the index is:
  Mild, between 5 and 15 per hour Moderate, between 15 and 30 per hour Severe, over than 30 per hour
Change in sleep quality | 60 days
  Sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI) questionnaire. This will be used to measure sleep quality over the last 60 days.The self-related questions include the assessment of seven different sleep domains : sleep quality, sleep latency , sleep duration , habitual sleep efficiency, sleep disturbances , use of sleeping medications , and daytime dysfunction .The seven components scores are then added to yield a global PSQI score in the range of zero to 21. The higher the score, the worse the sleep quality. A global score greater than five is diagnostic of poor sleep quality.
Change in sleepiness | 60 days
  Sleepiness will be assessed by the Epworth Sleepiness Scale (ESS).It will be used to measure daytime sleepiness .It can determine the chance of falling asleep in 8 different circumstances. ESS score can range from 0 to 24. A global score greater than ten is diagnostic of excessive daytime sleepiness .

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Laboratoire EFCR - CHU de Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided